CLINICAL TRIAL: NCT03955497
Title: Efficacy and Safety Research of Autologous Adipose-derived Mesenchymal Stem Cell Gel in the Treatment of Cartilage Damage in the Knee
Brief Title: Effectiveness of Autologous Adipose-derived Stem Cells in the Treatment of Knee Cartilage Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018023
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Knee Osteoarthritis; Cartilage Degeneration
Keywords: Knee Osteoarthritis; Stem Cell; Cartilage repair
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Adipose-derived Mesenchymal Stem Cell Gel (Experimental): The experimental group received intra-articular injection of Autologous Adipose-derived Mesenchymal Stem Cell Gel one month after operation.
  Interventions: Other: Autologous Adipose-derived Mesenchymal Stem Cell Gel; Procedure: Extraction of abdominal fat
- sodium hyaluronate (Placebo Comparator): The control group received intra-articular injection of sodium hyaluronate one month after operation.
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Other: Autologous Adipose-derived Mesenchymal Stem Cell Gel — The experimental group received intra-articular injection of Autologous Adipose-derived Mesenchymal Stem Cell Gel one month after operation.
  Arms: Autologous Adipose-derived Mesenchymal Stem Cell Gel
Drug: Sodium Hyaluronate — The control group received intra-articular injection of sodium hyaluronate one month after operation.
  Other Names: hyaluronic acid
  Arms: sodium hyaluronate
Procedure: Extraction of abdominal fat — In the experimental group, abdominal fat was extracted before operation to prepare Autologous Adipose-derived Mesenchymal Stem Cell Gel.
  Other Names: Fat extraction
  Arms: Autologous Adipose-derived Mesenchymal Stem Cell Gel

SUMMARY:
This study was aimed to evaluate the efficacy and safety of Autologous Adipose-derived Mesenchymal Stem Cell Gel combine with High tibial osteotomy therapy in the treatment of cartilage damage in the knee. Investigator believe that this method will enable patients to recover better knee function and more repair of knee cartilage.

DETAILED DESCRIPTION:
The patients who will underwent high tibial osteotomy were randomly divided into the experimental group and the control group. Abdominal fat extraction before operation in experimental group to prepare Adipose-derived Mesenchymal Stem Cell Gel, while the control group only underwent high tibial osteotomy. One month after operation, the experimental group was injected with Adipose-derived Mesenchymal Stem Cell Gel into the joint cavity, and the control group was injected with sodium hyaluronate in the joint cavity. Two groups of patients were followed up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years, male and female, patient can tolerate surgery;
* Clinical diagnosis of degenerative arthritis by Radiographic Criteria;
* Obviously extra-articular malformation;
* Good contralateral interventricular cartilage;
* Course of disease ≥ six months;
* There was no obvious abnormality in tumor marker detection,or patient was evaluated has not at the risk of cancer;
* Subjects who understand and sign the consent form for this study.

Exclusion Criteria:

* Acute joint injury;
* Patients with severe primary diseases, such as cardiovascular,cerebrovascular, liver, kidney and hematopoietic system, and psychosis;
* Cancer patients;
* Women who are pregnant or breast feeding,or allergic constitution patient;
* Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg, Anti-Hepatitis C virus -Ab), Hepatitis C (Anti-hepatitis C virus -Ab) and syphilis;
* Receive other open surgery related to knee operation within 6 months;
* Participation in another clinical trial;
* Failing to comply with the inclusion criteria, unwilling to comply with the research approach, or incomplete data affecting the curative effect or safety judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital for special surgery knee score postoperative 1 month | postoperative 1 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 3 month | postoperative 3 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 6 month | postoperative 6 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 12 month | postoperative 12 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 24 month | postoperative 24 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Hospital for special surgery knee score postoperative 36 month | postoperative 36 month
  Hospital for special surgery knee score is a knee function scoring system with a full score of 100. 0 means the loss of knee function, 100 means the best knee function, and the greater the value, the better knee function.
Visual Analogue Scale Postoperative Day 1 | Postoperative Day 1
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative Day 2 | Postoperative Day 2
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative Day 3 | Postoperative Day 3
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative Day 7 | Postoperative Day 7
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 1 month | Postoperative 1 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 3 month | Postoperative 3 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 6 month | Postoperative 6 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 12 month | Postoperative 12 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative Day One | Postoperative Day One
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 24 month | Postoperative 24month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Visual Analogue Scale Postoperative 36 month | Postoperative 36 month
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Evaluation of cartilage repair under MRI postoperative 12 month | Postoperative 12 month
  Recht criterion was used for grading articular cartilage injury of knee joint, including 0-IV grade, in which: 0 grade, normal articular cartilage, no obvious abnormal signal was found; 1 grade, the layered structure of cartilage disappeared, and there were focal low signal areas, but the surface was smooth; 2 grade, the surface of cartilage was irregular, the depth of cartilage injury was less than 50% cartilage thickness; 3 grade, the surface of cartilage was heavy. The degree of injury is irregular, the depth of injury is more than 50% of the thickness of cartilage or through the whole layer, but the surface of cartilage is not completely exfoliated; Grade IV, full-thickness cartilage defect, articular cartilage injury deep to the cortex, subchondral bone exposed.
Evaluation of cartilage repair under MRI postoperative 24 month | Postoperative 24 month
  Recht criterion was used for grading articular cartilage injury of knee joint, including 0-IV grade, in which: 0 grade, normal articular cartilage, no obvious abnormal signal was found; 1 grade, the layered structure of cartilage disappeared, and there were focal low signal areas, but the surface was smooth; 2 grade, the surface of cartilage was irregular, the depth of cartilage injury was less than 50% cartilage thickness; 3 grade, the surface of cartilage was heavy. The degree of injury is irregular, the depth of injury is more than 50% of the thickness of cartilage or through the whole layer, but the surface of cartilage is not completely exfoliated; Grade IV, full-thickness cartilage defect, articular cartilage injury deep to the cortex, subchondral bone exposed.
Evaluation of cartilage repair under MRI postoperative 36 month | Postoperative 36 month
  Recht criterion was used for grading articular cartilage injury of knee joint, including 0-IV grade, in which: 0 grade, normal articular cartilage, no obvious abnormal signal was found; 1 grade, the layered structure of cartilage disappeared, and there were focal low signal areas, but the surface was smooth; 2 grade, the surface of cartilage was irregular, the depth of cartilage injury was less than 50% cartilage thickness; 3 grade, the surface of cartilage was heavy. The degree of injury is irregular, the depth of injury is more than 50% of the thickness of cartilage or through the whole layer, but the surface of cartilage is not completely exfoliated; Grade IV, full-thickness cartilage defect, articular cartilage injury deep to the cortex, subchondral bone exposed.
Degree of meniscus injury under MRI postoperative 12 month | postoperative 12 month
  Stoller's criteria were used in the classification of meniscal injuries, including 0-3 grades, in which: 0 grade, the shape of meniscus was regular, complete and even low signal; 1 grade, focal ellipse or circular high signal appeared in the meniscus, which did not extend to the articular surface and margin of the meniscus; 2 grade, the meniscus showed horizontal linear high signal extending to the articular margin of the meniscus.
  But it did not exceed the articular surface; in grade III, the shape of meniscus was irregular and incomplete. Irregular or linear high signal appeared in the meniscus and extended to the articular surface of meniscus. The grade I and II symptoms of meniscus injury were mild, suggesting meniscus degeneration, and grade III suggesting meniscus tear.
Degree of meniscus injury under MRI postoperative 24 month | postoperative 24 month
  Stoller's criteria were used in the classification of meniscal injuries, including 0-3 grades, in which: 0 grade, the shape of meniscus was regular, complete and even low signal; 1 grade, focal ellipse or circular high signal appeared in the meniscus, which did not extend to the articular surface and margin of the meniscus; 2 grade, the meniscus showed horizontal linear high signal extending to the articular margin of the meniscus.
  But it did not exceed the articular surface; in grade III, the shape of meniscus was irregular and incomplete. Irregular or linear high signal appeared in the meniscus and extended to the articular surface of meniscus. The grade I and II symptoms of meniscus injury were mild, suggesting meniscus degeneration, and grade III suggesting meniscus tear.
Degree of meniscus injury under MRI postoperative 36 month | postoperative 36 month
  Stoller's criteria were used in the classification of meniscal injuries, including 0-3 grades, in which: 0 grade, the shape of meniscus was regular, complete and even low signal; 1 grade, focal ellipse or circular high signal appeared in the meniscus, which did not extend to the articular surface and margin of the meniscus; 2 grade, the meniscus showed horizontal linear high signal extending to the articular margin of the meniscus.
  But it did not exceed the articular surface; in grade III, the shape of meniscus was irregular and incomplete. Irregular or linear high signal appeared in the meniscus and extended to the articular surface of meniscus. The grade I and II symptoms of meniscus injury were mild, suggesting meniscus degeneration, and grade III suggesting meniscus tear.
Evaluation of cartilage repair under arthroscope postoperative 12 month | postoperative 12 month
  The arthroscopic classification of knee joint cartilage injury refers to the classification criteria formulated by the International Association of Cartilage Repair, which includes 0-IV grades, of which: 0 grade is normal articular cartilage; 1 grade is the surface injury of cartilage with soft edema on the surface, with only small cracks and intact structure; 2 grade is partial cartilage injury, which extends downward from the surface, but the depth of injury is less than 50% cartilage thickness. Grade III, deep articular injury, injury depth > 50% cartilage thickness or through the whole layer; Grade IV, deep articular cartilage injury to the bone cortex, full-thickness cartilage defect, subchondral bone exposure.
Degree of meniscus injury under arthroscope postoperative 12 month | postoperative 12 month
  The degree of meniscus injury under arthroscopy was classified into three grades, including normal, degenerative and tear.

SECONDARY OUTCOMES:
Squatting to Standing Time postoperative 1 month | postoperative 1 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 3 month | postoperative 3 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 6 month | postoperative 6 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 12 month | postoperative 12 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 24 month | postoperative 24 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.
Squatting to Standing Time postoperative 36 month | postoperative 36 month
  The patient squatted on the floor and then stood up completely for five consecutive times, recording the time required.

CONTACTS AND LOCATIONS:
Overall Officials: Peilai Liu, MD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The acquisition of individual participant data needs the consent of Peilai Liu, the person in charge.

REFERENCES:
- [Background] Yu D, Xu J, Liu F, Wang X, Mao Y, Zhu Z. Subchondral bone changes and the impacts on joint pain and articular cartilage degeneration in osteoarthritis. Clin Exp Rheumatol. 2016 Sep-Oct;34(5):929-934. Epub 2016 Aug 31. PMID 27606839
- [Background] Wilusz RE, Sanchez-Adams J, Guilak F. The structure and function of the pericellular matrix of articular cartilage. Matrix Biol. 2014 Oct;39:25-32. doi: 10.1016/j.matbio.2014.08.009. Epub 2014 Aug 27. PMID 25172825
- [Background] Baer PC, Geiger H. Adipose-derived mesenchymal stromal/stem cells: tissue localization, characterization, and heterogeneity. Stem Cells Int. 2012;2012:812693. doi: 10.1155/2012/812693. Epub 2012 Apr 12. PMID 22577397
- [Background] Chareancholvanich K, Pornrattanamaneewong C, Narkbunnam R. Increased cartilage volume after injection of hyaluronic acid in osteoarthritis knee patients who underwent high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2014 Jun;22(6):1415-23. doi: 10.1007/s00167-013-2735-1. Epub 2013 Oct 27. PMID 24162762